CLINICAL TRIAL: NCT00339963
Title: Expression of the Genome in Lymphoid Malignancies
Brief Title: Genome Expression in Lymphoma, Leukemia and Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Lymphoma/Leukemia Molecular Profiling Project (LLMPP) (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902042; 02-C-N042
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-03-13

CONDITIONS: Leukemia; Multiple Myeloma; Hodgkin Lymphoma; Lymphoma, Non-Hodgkin
Keywords: Microarray; Lymphoma; Gene Expression; Molecular Diagnosis; Prognosis; Natural History; Leukemia; Myeloma; Lymphoid Malignancy
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will use genomics-based technology, such as DNA microarrays, to more precisely diagnose subsets of lymphoma, leukemia and multiple myeloma patients. There have been many attempts to classify lymphoid cancers in ways that will be useful for clinical diagnosis and treatment. Although broad diagnostic categories have been reliably defined, patients within each category have distinct clinical courses, suggesting that these classifications could be further divided into molecular (genetic) subtypes. For example, 40 percent of patients with diffuse large B-cell lymphoma achieve long-term disease remissions following combination chemotherapy and are apparently cured, whereas the remaining 60 percent die from the disease. Similarly, some patients with follicular lymphoma develop aggressive disease within a few years of diagnosis, while others have stable disease over 10 to 20 years. Although the distinctions in clinical course of these diseases are recognized, there are no studies to determine the molecular (genetic) basis for this variability. This study will try to define new molecular diagnostic categories in these diseases and correlate them with clinical features, including treatment response, disease remission and overall survival following chemotherapy.

This retrospective study will use clinical data and tissue samples from participating centers in the Lymphoma/Leukemia Molecular Profiling Project LLMPP). New patients will not be recruited for this study.

Biopsy materials, including fresh frozen or OTC-embedded lymphoma biopsy material, viably frozen samples of peripheral blood cells from leukemia patients, and viably frozen samples of bone marrow aspirates from multiple myeloma patients will be collected from pathologists participating in the LLMPP. RNA and genomic DNA will be extracted from the tumor samples. A variety of technologies will be used to characterize the genome of the cancer cells, including lymphochip microarrays for array-based comparative genomic hybridization; Southern blotting and PCR for translocation of genes previously implicated in these malignancies; and PCR and DNA sequencing methods for analyzing base changes in the genome of the cancer cells. Clinical information from the initial diagnosis to disease relapse will be taken from existing databases and/or patient charts. Gene expression will be correlated with the clinical data. If a small number of genes is found to strongly predict clinical outcome, quantitative RT-PCR assays using the Taqman technology may be developed as an alternative to DNA microarray analysis.

...

DETAILED DESCRIPTION:
Current diagnosis of the lymphoid malignancies relies upon the morphological appearance of the cancer cells supplemented by a few molecular markers. Within a diagnostic category, the clinical courses and responses of patients to therapy are variable, suggesting that the existing diagnostic categories may harbor more than one disease entity. Recent genomic technologies allow a comprehensive molecular analysis of the expression of the genome in cancer cells. DNA microarray analysis of gene expression in lymphomas revealed distinct molecular subtypes of diffuse large B-cell lymphoma and these new molecularly-defined lymphoma subtypes had divergent clinical outcomes. To extend our genomic analysis to all lymphoid malignancies, we have formed a consortium of cooperating institutions termed the Lymphoma/Leukemia Molecular Profiling Project (LLMPP). The clinical centers participating in the LLMPP will send de-identified lymphoma, leukemia and multiple myeloma samples to the NCI for gene expression profiling, array-based comparative genomic hybridization and cancer gene resequencing. An additional site, The National Cancer Center Singapore, will send de-identified samples of tumor tissue from patients with lymphoma.

Objective:

Assess gene expression on a genomic scale in lymphoma, leukemia and multiple myeloma samples and its relationship to somatic genetic alterations.

Eligibility:

Diagnosis of lymphoid malignancy at one of the LLMPP participating institutions, including specimens originating at other clinical sites and submitted to LLMPP participating sites or The National Cancer Center Singapore.

Design:

This is an entirely retrospective study. All tumor biopsies containing malignant cells to be analyzed were obtained previously from patients diagnosed and/or treated at one of the institutions participating in the LLMPP or at The National Cancer Center Singapore.

Clinical data will also be sent for the patients in this study for the purpose of correlating gene expression measurements with clinical outcome. The goals of this effort are to define new molecular diagnostic categories in these diseases that are clinically relevant and to gain new insight into the molecular pathways that are active in these malignancies.

The home institutions providing clinical data and tissue samples have obtained local approval by their clinical research committees for this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of lymphoid malignancy at one of the LLMPP participating institutions, including specimens originating at other clinical sites and submitted to LLMPP participating sites or National Cancer Center Singapore.

Informed consent for research studies performed on biopsy material or waiver of the requirement for informed consent by the clinical research review boards at the LLMPP institutions or National Cancer Center Singapore.

Sufficient frozen biopsy and/or FFPE material from initial biopsy and/or biopsies at relapse of disease to obtain adequate RNA and DNA for gene expression profiling and analysis of genomic alterations in the malignant cells.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed and/or treated at one of the institutions participating in the LLMPP or at The National Cancer Center Singapore.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1340 (Actual)
Dates: Start 2001-11-09

PRIMARY OUTCOMES:
Gene expression on a genomic scale in lymphoma, leukemia and multiple myeloma samples. | Every year
  Define new molecular diagnostic categories in these diseases that are clinically relevant and to gain new insight into the molecular pathways that are active in these malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Staudt, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gascoyne RD, Adomat SA, Krajewski S, Krajewska M, Horsman DE, Tolcher AW, O'Reilly SE, Hoskins P, Coldman AJ, Reed JC, Connors JM. Prognostic significance of Bcl-2 protein expression and Bcl-2 gene rearrangement in diffuse aggressive non-Hodgkin's lymphoma. Blood. 1997 Jul 1;90(1):244-51. PMID 9207459
- [Background] Vose JM. Current approaches to the management of non-Hodgkin's lymphoma. Semin Oncol. 1998 Aug;25(4):483-91. PMID 9728598
- [Background] Harris NL, Jaffe ES, Stein H, Banks PM, Chan JK, Cleary ML, Delsol G, De Wolf-Peeters C, Falini B, Gatter KC, et al. A revised European-American classification of lymphoid neoplasms: a proposal from the International Lymphoma Study Group. Blood. 1994 Sep 1;84(5):1361-92. No abstract available. PMID 8068936